CLINICAL TRIAL: NCT03964805
Title: Impact of Low Versus Atmospheric Oxygen Tension on Human Embryo Development : A Prospective Randomized Study
Brief Title: Oxygen Tension on Human Embryonic Development
Acronym: EmbryOx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A02019-40
Record Dates: First submitted 2019-05-14; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-04

CONDITIONS: Infertility; Embryo Culture; Hypoxia
Keywords: Embryo culture; oxygen tension,; embryo quality,; extended culture
MeSH Terms: conditions — Infertility; Hypoxia | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): Embryo culture at 20% O2
  Interventions: Other: 20% oxygen
- group B (Active Comparator): Embryo culture at 5% O2
  Interventions: Other: 5% oxygen
- group C (Active Comparator): Embryo culture at 5% O2 and at 20% O2
  Interventions: Other: 20 % and 5 % oxygen

INTERVENTIONS:
Other: 20% oxygen — culture excusively at 20% O2 (Day 0 to Day 6)
  Other Names: culture at 20% O2
  Arms: group A
Other: 5% oxygen — culture excusively at 5% O2 (Day 0 to Day 6)
  Other Names: culture at 5% O2
  Arms: group B
Other: 20 % and 5 % oxygen — culture at 5% from Day 0 to Day 3, then at 20% from Day 3 to Day 6)
  Other Names: culture at 20 % and at 5%O2
  Arms: group C

SUMMARY:
In mammals, uterine environment is at low oxygen concentration (2-8% O2). Thus, human embryo culture under low O2 tension (5%) is now recommended by European Society of Human Reproduction and Embryology (ESHRE) revised guidelines for good practices in in vitro fertilization (IVF) labs. Indeed, hypoxia seems to improve embryo quality at cleavage and blastocyst stages, presumably by reducing damages of oxidative stress (OS). Nevertheless, recent meta-analyses concluded only with a low evidence to a superiority of hypoxia on IVF/ICSI outcomes. Furthermore, a study on mouse embryos suggested a negative impact of OS only at cleavage stage. The aim of the present prospective randomized study was to investigate this hypothesis for the first time in human embryos.

DETAILED DESCRIPTION:
In mammals, uterine environment is at low oxygen tension, between 2 and 8% O2 . However, most IVF labs perform embryo culture at atmospheric tension (around 20% O2). Several randomized studies in human embryos have reported the superiority of hypoxia (5%) in terms of embryo quality and blastulation rates. This fact might be explained by a more physiological environment, probably inducing a decrease in oxidative stress (OS), which has a harmful impact on embryo development. Other studies have also suggested that before compaction, OS damages might be irreversible.

Wale et Gardner have investigated this impact of oxygen tension on mouse embryo development, by comparing four culture conditions: (i) group 1: culture exclusively at 5% O2 ; (ii) group 2: culture at 5% from Day 0 to Day 2, then at 20% from Day 2 to Day 4; (iii) group 3: at 20% then at 5% from Day 2; (iv) and group 4: culture exclusively at 20% Interestingly, no difference in terms of blastulation had been reported between groups 1 and 2, suggesting the OS might impact only at cleavage stage, and that switching culture under atmospheric conditions from Day 2/3 might not influence embryo development thereafter.

Hence, all those investigations suggest that embryo culture using trigas incubators (5% O2, 6% CO2 and 89% N2) would be preferable. However, this system is very expensive, notably due to a high N2 consumption, and requires a more complicated logistics (e.g. N2 levels monitoring). Yet, Wale and Gardner's results imply that sequential culture conditions (trigas from Day 0 to Day 2/3, then conventional incubator at 20% O2 until blastocyst stage) could be an valuable option, reducing the costs and, essentially, without any detrimental impact on embryo development.

The present study has two main objectives: (i) to confirm the improvement in embryo quality under low oxygen tension and (ii) to demonstrate the negative impact of OS only at cleavage stage in human embryos, as assumed by Wale and Gardner. For that purpose, we designed an original prospective randomized study comparing three culture conditions: (i) culture excusively at 20% O2 (Day 0 to Day 6) (Group A); (ii) culture exclusively at 5% O2 (Day 0 to Day 6) (Group B); (iii) culture at 5% from Day 0 to Day 3, then at 20% from Day 3 to Day 6) (Group C). Inclusion criteria and outcome measures are detailed in the following sections.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 39 years
* IVF / ICSI Attempt with Ejaculated Sperm Sperm (Fresh or Frozen)
* At least 8 oocytes retrieved in total
* Good understanding of the protocol by the patient
* Informed and consentment signed of the couple

Exclusion Criteria:

* - Hydrosalpinx

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 773 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Embryo quality at Day 2 between groups A and B. | Day 2
  Embryo morphology is qualified as the number of blastomeres, degree of cytoplasmic fragmentation, regularity of the cells and presence/absence of multinucleated blastomeres. Day 2 top-quality embryos are defined as 4 regular blastomeres, <20% cytoplasmic fragmentation, no multinucleations.mbryos are defined as 4/8 regular blastomeres, <20% cytoplasmic fragmentation, no multinucleations.
Embryo quality at Day 3 between groups A and B. | Day 3
  Embryo morphology is qualified as the number of blastomeres, degree of cytoplasmic fragmentation, regularity of the cells and presence/absence of multinucleated blastomeres. Day 3 top-quality embryos are defined as 8 regular blastomeres, <20% cytoplasmic fragmentation, no multinucleations.
Embryo quality at blastocyst stage (Day 5) between groups A, B and C. | Day 5
  Blastocyst morphology is assessed according to Gardner and Schoolcraft's classification: degree of blastocele expansion (graded from B1 to B6), inner cell mass and trophectoderm morphology (both graded A, B or C). Day 5 top quality blastocyst are defined as ≥B4AA/AB/BA.
Embryo quality at blastocyst stage (Day 6) between groups A, B and C. | Day 6
  Blastocyst morphology is assessed according to Gardner and Schoolcraft's classification: degree of blastocele expansion (graded from B1 to B6), inner cell mass and trophectoderm morphology (both graded A, B or C). Day 5 top quality blastocyst are defined as ≥B4AA/AB/BA.

SECONDARY OUTCOMES:
Fertilization rate | Days 1
  Percentage of oocytes fertilized per oocyte inseminated, assessed at Day 1
Early cleavage rate | 25 hours after insemination
  Percentage of embryos at the 2-cell stage per oocyte fertilized, assessed 25 hours after insemination
Useable embryo rate | Days 2/3; 5/6
  Percentage of embryos transferred and/or frozen per embryo
Implantation rate | 4-5 weeks after transfer
  Number of gestational sacs with fetal heart beat detected per embryo transferred
Clinical pregnancy rate | 4-5 weeks after transfer
  Percentage of pregnancies diagnosed by ultrasonographic visualization of at least one gestational sac with fetal heart beat per embryo transfer
Miscarriage rate | 4-5 weeks after transfer

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Sifer, Principal Investigator — AP-HP_Hôpital Jean Verdier

REFERENCES:
- [Background] Ciray HN, Aksoy T, Yaramanci K, Karayaka I, Bahceci M. In vitro culture under physiologic oxygen concentration improves blastocyst yield and quality: a prospective randomized survey on sibling oocytes. Fertil Steril. 2009 Apr;91(4 Suppl):1459-61. doi: 10.1016/j.fertnstert.2008.07.1707. Epub 2008 Aug 22. PMID 18722608
- [Background] Fischer B, Bavister BD. Oxygen tension in the oviduct and uterus of rhesus monkeys, hamsters and rabbits. J Reprod Fertil. 1993 Nov;99(2):673-9. doi: 10.1530/jrf.0.0990673. PMID 8107053
- [Background] Guo N, Li Y, Ai J, Gu L, Chen W, Liu Q. Two different concentrations of oxygen for culturing precompaction stage embryos on human embryo development competence: a prospective randomized sibling-oocyte study. Int J Clin Exp Pathol. 2014 Aug 15;7(9):6191-8. eCollection 2014. PMID 25337269
- [Background] Kasterstein E, Strassburger D, Komarovsky D, Bern O, Komsky A, Raziel A, Friedler S, Ron-El R. The effect of two distinct levels of oxygen concentration on embryo development in a sibling oocyte study. J Assist Reprod Genet. 2013 Aug;30(8):1073-9. doi: 10.1007/s10815-013-0032-z. Epub 2013 Jul 9. PMID 23835722
- [Background] Kea B, Gebhardt J, Watt J, Westphal LM, Lathi RB, Milki AA, Behr B. Effect of reduced oxygen concentrations on the outcome of in vitro fertilization. Fertil Steril. 2007 Jan;87(1):213-6. doi: 10.1016/j.fertnstert.2006.05.066. Epub 2006 Nov 1. PMID 17081523
- [Background] Kirkegaard K, Hindkjaer JJ, Ingerslev HJ. Effect of oxygen concentration on human embryo development evaluated by time-lapse monitoring. Fertil Steril. 2013 Mar 1;99(3):738-744.e4. doi: 10.1016/j.fertnstert.2012.11.028. Epub 2012 Dec 11. PMID 23245683
- [Background] Kovacic B, Vlaisavljevic V. Influence of atmospheric versus reduced oxygen concentration on development of human blastocysts in vitro: a prospective study on sibling oocytes. Reprod Biomed Online. 2008 Aug;17(2):229-36. doi: 10.1016/s1472-6483(10)60199-x. PMID 18681997
- [Background] Waldenstrom U, Engstrom AB, Hellberg D, Nilsson S. Low-oxygen compared with high-oxygen atmosphere in blastocyst culture, a prospective randomized study. Fertil Steril. 2009 Jun;91(6):2461-5. doi: 10.1016/j.fertnstert.2008.03.051. Epub 2008 Jun 12. PMID 18554591
- [Background] Wale PL, Gardner DK. Time-lapse analysis of mouse embryo development in oxygen gradients. Reprod Biomed Online. 2010 Sep;21(3):402-10. doi: 10.1016/j.rbmo.2010.04.028. Epub 2010 Aug 5. PMID 20691637
- [Background] Wale PL, Gardner DK. The effects of chemical and physical factors on mammalian embryo culture and their importance for the practice of assisted human reproduction. Hum Reprod Update. 2016 Jan-Feb;22(1):2-22. doi: 10.1093/humupd/dmv034. Epub 2015 Jul 22. PMID 26207016